CLINICAL TRIAL: NCT05515198
Title: Empowering Women and Providers for Improved Care of Urinary Incontinence (UI) [EMPOWER Study]
Brief Title: Improving Care for Women With Urinary Incontinence (EMPOWER)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Adonis Hijaz, MD, Vice Chair of Academics and Research for the Urology Institute, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20211420
Record Dates: First submitted 2022-08-23; First posted 2022-08-25 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Urinary Incontinence
Keywords: women; female; urinary incontinence; empowering; EMPOWER; providers; bladder leakage; incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Patient Education as Topic; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Patient Education
  Interventions: Other: Patient Education
- Arm 2 (Experimental): Patient Education + Nurse Navigation
  Interventions: Other: Patient Education; Other: Nurse Navigation
- Arm 3 (Experimental): Patient Education + Nurse Navigation + ChatBot
  Interventions: Other: Patient Education; Other: Nurse Navigation; Other: ChatBot

INTERVENTIONS:
Other: Patient Education — Patients will be provided educational opportunities.
  Other Names: Education
Other: Nurse Navigation — A nurse navigator will work with the participants to help them navigate the care pathway. The navigator will provide education and recommendations for treatment options.
  Arms: Arm 2; Arm 3
Other: ChatBot — A ChatBot will allow participants to directly and privately communicate through a smartphone (or other device) with an artificial intelligence-driven ChatBot, also known as a "conversational agent," that will provide education and encouragement to manage their symptoms.
  Other Names: Behavioral/exercise via chatbot
  Arms: Arm 3

SUMMARY:
The overall goal is to improve diagnosis and non-operative management of urinary incontinence in women.

DETAILED DESCRIPTION:
In the study, patients will be screened in primary care offices for symptoms of urinary incontinence. Women with positive screening results will be asked if they are interested in participating in an implementation study where women will be assigned to one of the three following groups:

1. Usual Care plus Patient Educational Opportunities - The patient's urinary incontinence will be managed using standard of care treatment by the patient's primary care provider. Patients will be offered educational opportunities about urinary incontinence.
2. Nurse Navigation - Along with the treatment described for "Usual Care plus Patient Educational Opportunities," a nurse navigator will work with the patient to implement behavioral changes and provide education and physical therapy options. In addition, the navigator will be available to answer the patient's questions in a timely fashion and help the patient move through the care pathway.
3. Nurse Navigation and ChatBot - Along with the treatment described for "Usual Care plus Patient Educational Opportunities" and "Nurse Navigation," this group will include a ChatBot feature which will allow a patient to directly and privately communicate with an artificial intelligence-driven ChatBot, also known as a "conversational agent," that will provide education and help the patient navigate the care pathway.

All participants will complete questionnaires throughout their enrollment and data will be collected from medical records. The study team will analyze the data at six months after the original appointment/study enrollment, assess adherence to therapy and how the therapy impacted the outcomes the team hopes to improve, such as improvement in symptoms. The study will be implemented over three subsequent time periods called Wave 1, Wave 2 and Wave 3 with primary care practices from two geographic regions being involved in each wave (6 regions total). Participants in Wave 1 will be followed for a total of 18 months, while participants in Wave 2 will be followed for a total of 12 months, and participants in Wave 3 will be followed for 6 months. Primary care providers at all participating practices will be offered educational opportunities related to urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Female patient having a primary care provider visit at University Hospitals (UH) Cleveland Primary Care Institute (PCI)
2. ≥ 18 years old
3. Scores 1 or higher on the International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-SF)

Exclusion Criteria:

None

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females only
Enrollment: 400 (Actual)
Dates: Start 2022-09-06 (Actual); Primary Completion 2024-12-23 (Actual); Study Completion 2024-12-23 (Actual)

PRIMARY OUTCOMES:
Change in patients' UI symptoms as measured by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | Baseline and Months 2 and 6 (all Waves)
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) assess frequency, severity and impact on quality of life (QoL) of patients' urinary incontinence symptoms. The result of the ICIQ-UI SF is a composite score ranging from 0 to 21, with higher scores indicating more severe incontinence.
Patients' UI symptoms as measured by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | 12 months (Waves 1 and 2)
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) assess frequency, severity and impact on quality of life (QoL) of patients' urinary incontinence symptoms. The result of the ICIQ-UI SF is a composite score ranging from 0 to 21, with higher scores indicating more severe incontinence.
Patients' UI symptoms as measured by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) | 18 months (Wave 1)
  The International Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-UI SF) assess frequency, severity and impact on quality of life (QoL) of patients' urinary incontinence symptoms. The result of the ICIQ-UI SF is a composite score ranging from 0 to 21, with higher scores indicating more severe incontinence.

SECONDARY OUTCOMES:
Change in patients' perceived self-efficacy for UI communication as measured by the PEPPI | Baseline and Months 2 and 6 (all Waves)
  Patients' perceived confidence in their ability to communicate their health concerns around UI will be assessed by the Patient-Perceived Self-Efficacy in Patient-Physician Interactions (PEPPI) Questionnaire modified for UI. The PEPPI total score ranges from 0 to 50, with higher scores indicating greater self-efficacy.
Patients' perceived self-efficacy for UI communication as measured by the PEPPI | 12 months (Waves 1 and 2)
  Patients' perceived confidence in their ability to communicate their health concerns around UI will be assessed by the Patient- Perceived Self-Efficacy in Patient-Physician Interactions (PEPPI) Questionnaire modified for UI. The PEPPI total score ranges from 0 to 50, with higher scores indicating greater self-efficacy.
Patients' perceived self-efficacy for UI communication as measured by the PEPPI | 18 months (Wave 1)
  Patients' perceived confidence in their ability to communicate their health concerns around UI will be assessed by the Patient- Perceived Self-Efficacy in Patient-Physician Interactions (PEPPI) Questionnaire modified for UI. The PEPPI total score ranges from 0 to 50, with higher scores indicating greater self-efficacy.
Change in patient empowerment as measured by a patient survey | Baseline and Months 2 and 6 (all Waves)
  Patient empowerment will be measured by a patient survey to measure with percentage of patients answering yes to speaking with their provider about UI.
Change in overactive bladder symptom severity as measured by the OABSS | Baseline and Months 2 and 6 (all Waves)
  Patients' overactive bladder symptom severity will be assessed by the Overactive Bladder Symptom Score (OABSS). The OABSS total score ranges from 0 to 15, with higher scores indicating more severe symptoms.
Overactive bladder symptom severity as measured by the OABSS | 12 months (Waves 1 and 2)
  Patients' overactive bladder symptom severity will be assessed by the Overactive Bladder Symptom Score (OABSS). The OABSS total score ranges from 0 to 15, with higher scores indicating more severe symptoms.
Overactive bladder symptom severity as measured by the OABSS | 18 months (Wave 1)
  Overactive bladder symptom severity will be assessed by the Overactive Bladder Symptom Score (OABSS). The OABSS total score ranges from 0 to 15, with higher scores indicating more severe symptoms.
Change in urinary symptoms as measured by the UDI-6 | Baseline and Months 2 and 6 (all Waves)
  How bothersome a patient's urinary symptoms are will be assessed by the Urinary Distress Inventory (UDI-6). The UDI-6 total score ranges from 0 to 100, with higher scores indicating more bothersome symptoms.
Urinary symptoms as measured by the UDI-6 | 12 months (Waves 1 and 2)
  How bothersome a patient's urinary symptoms are will be assessed by the Urinary Distress Inventory (UDI-6). The UDI-6 total score ranges from 0 to 100, with higher scores indicating more bothersome symptoms.
Urinary symptoms as measured by the UDI-6 | 18 months (Wave 1)
  How bothersome a patient's urinary symptoms are will be assessed by the Urinary Distress Inventory (UDI-6). The UDI-6 total score ranges from 0 to 100, with higher scores indicating more bothersome symptoms.
Change in impact of UI on patients' quality of life as measured by the ICIQ-LUTSqol | Baseline and Months 2 and 6 (all Waves)
  The impact of urinary incontinence on quality of life will be assessed by the Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol total score ranges from 19 to 76, with higher scores indicating increased impact on quality of life.
Impact of UI on patients' quality of life as measured by the ICIQ-LUTSqol | 12 months (Waves 1 and 2)
  The impact of urinary incontinence on quality of life will be assessed by the Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol total score ranges from 19 to 76, with higher scores indicating increased impact on quality of life.
Impact of UI on patients' quality of life as measured by the ICIQ-LUTSqol | 18 months (Wave 1)
  The impact of urinary incontinence on quality of life will be assessed by the Incontinence Questionnaire Lower Urinary Tract Symptoms Quality of Life Module (ICIQ-LUTSqol). The ICIQ-LUTSqol total score ranges from 19 to 76, with higher scores indicating increased impact on quality of life.
Change in patients' perceived symptom improvement as measured by the PGI-I | Months 2 and 6 (all Waves)
  Patients' perceived improvement in UI symptoms will be assessed with the Patient Global Impression of Improvement (PGI-I). PGI-I measures improvement on a scale of 1 "very much better" to 7 "very much worse."
Patients' perceived symptom improvement as measured by the PGI-I | 12 months (Waves 1 and 2)
  Patients' perceived improvement in UI symptoms will be assessed with the Patient Global Impression of Improvement (PGI-I). PGI-I measures improvement on a scale of 1 "very much better" to 7 "very much worse."
Patients' perceived symptom improvement as measured by the PGI-I | 18 months (Wave 1)
  Patients' perceived improvement in UI symptoms will be assessed with the Patient Global Impression of Improvement (PGI-I). PGI-I measures improvement on a scale of 1 "very much better" to 7 "very much worse."
Number of practices that maintain a UI management intervention as measured by the practice survey | 1 month post completion of each Wave's enrollment period
  Maintenance of UI management intervention will be assessed by practice survey with indication of continuation for each intervention component.
Number of practices that implement a UI point person as measured by the practice survey | 1 month post completion of each Wave's enrollment period
  Implementation of a UI point person will be measured as a percentage of sites answer yes on practice survey.

CONTACTS AND LOCATIONS:
Overall Officials: Adonis Hijaz, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Goutham Rao, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following publication.
Access Criteria: Researchers who provide a methodologically sound proposal may use the data for any purpose.